CLINICAL TRIAL: NCT01943136
Title: The Efficacy and Safety of Topical Papaya (Carica Papaya) Leaf Extract 1% Ointment Versus Mupirocin 2% Ointment in the Treatment of Limited Impetigo: a Randomized, Double-blind, Controlled Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philippine Dermatological Society (Network)
Collaborators: St. Luke's Medical Center (Other)
Responsible Party: Principal Investigator, Pearl Weena Marie Sabido, Dr., Philippine Dermatological Society
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Papaya for impetigo
Record Dates: First submitted 2013-08-30; First posted 2013-09-16 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Impetigo
Keywords: impetigo; papaya extract ointment
MeSH Terms: conditions — Impetigo | interventions — Mupirocin; Ointments

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- papaya 1% extract ointment (Experimental): papaya 1% extract ointment twice a day for 1 week
  Interventions: Drug: papaya 1% extract ointment
- mupirocin 2% ointment (Active Comparator): mupirocin 2% ointment twice a day for 1 week
  Interventions: Drug: mupirocin 2% ointment

INTERVENTIONS:
Drug: papaya 1% extract ointment
  Arms: papaya 1% extract ointment
Drug: mupirocin 2% ointment
  Arms: mupirocin 2% ointment

SUMMARY:
This study will be an investigator-blinded, patient-blinded, assessor-blinded, parallel-group, randomized clinical trial. It aims to evaluate the efficacy of one-week twice-daily application of topical papaya leaf extract ointment compared to mupirocin ointment in achieving clinical cure among patients with impetigo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Filipino patients aged 1 year and above with primary impetigo, limited to less than or equal to 1% BSA, and involving only one body area

Exclusion Criteria:

* Extensive impetigo (>1% BSA), affecting more than one body area
* Systemic involvement (lymphadenopathy, fever, sepsis)
* Chronic comorbidities like diabetes mellitus, malignancy, chronic venous insufficiency
* Concurrent immunosuppressive therapy
* Patients ≤ 1 year
* Pregnant & lactating patients

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Clinical clearance after 1 week of treatment | 1 week

SECONDARY OUTCOMES:
time to clinical clearance | 1 week
score in the 6-point grading system | 1 week
  The 6-point grading system will assess clinical response based on each of the following six paramaters. One point will be assigned for each of the following parameters present in a patient, with the maximum possible score on this grading system being 6. A patient need not satisfy all six parameters. A decrease in score on this grading system compared to baseline will indicate clinical improvement, while an increase in score will indicate clinical worsening.
  * erythema
  * edema
  * vesiculation
  * pustulation
  * crusting
  * scaling
change in size of lesion compared to baseline | 1 week
presence or absence of recurrence on any part of the body 2 weeks after starting treatment | 1 week
presence or absence of adverse events during treatment | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Mia Angela C Verzosa, MD, Study Director — St. Luke's Medical Center; Pearl Weena Marie E Sabido, MD, Principal Investigator — St. Luke's Medical Center; Janine L. Quijano, MD, Principal Investigator — St. Luke's Medical Center
Locations (1):
- St. Luke's Medical Center, Quezon City, NCR, Philippines

REFERENCES:
- [Background] Koning S, van der Sande R, Verhagen AP, van Suijlekom-Smit LW, Morris AD, Butler CC, Berger M, van der Wouden JC. Interventions for impetigo. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD003261. doi: 10.1002/14651858.CD003261.pub3. PMID 22258953
- [Background] Craft N, Lee PK, Zipoli MT, Weinberg AN, Swartz MN, Johnson RA. "Superficial cutaneous infections and pyodermas." Ftizpatrick's Dermatology in General Medicine, 7th ed. Ed. Wolff K, et al. USA: McGraw-Hill Companies, 2008. 1694-1709.
- [Background] Woodford N, Livermore DM. Infections caused by Gram-positive bacteria: a review of the global challenge. J Infect. 2009 Sep;59 Suppl 1:S4-16. doi: 10.1016/S0163-4453(09)60003-7. PMID 19766888
- [Background] Witte W, Cuny C, Klare I, Nubel U, Strommenger B, Werner G. Emergence and spread of antibiotic-resistant Gram-positive bacterial pathogens. Int J Med Microbiol. 2008 Jul;298(5-6):365-77. doi: 10.1016/j.ijmm.2007.10.005. Epub 2008 Mar 5. PMID 18325835
- [Background] Pineda-Rebong AM, Tan JGB. Comparison of 2% oxytetracycline ointment with 2% mupirocin ointment and 2% sodium fusidate ointment in the treatment of impetigo in children: a preliminary report. J Phil Dermatol Soc 2011 May;20(1):21-4.
- [Background] Martin KW, Ernst E. Herbal medicines for treatment of bacterial infections: a review of controlled clinical trials. J Antimicrob Chemother. 2003 Feb;51(2):241-6. doi: 10.1093/jac/dkg087. PMID 12562687
- [Background] Anibijuwon II, Udeze AO. Antimicrobial activity of Carica papaya (pawpaw) leaf on some pathogenic organisms of clinical origin from south-western Nigeria. Ethnobotanical Leaflets 2009;13:850-64.
- [Background] Pieper B, Caliri MH. Nontraditional wound care: A review of the evidence for the use of sugar, papaya/papain, and fatty acids. J Wound Ostomy Continence Nurs. 2003 Jul;30(4):175-83. doi: 10.1067/mjw.2003.131. PMID 12851592
- [Background] Hewitt H, Whittle S, Lopez S, Bailey E, Weaver S. Topical use of papaya in chronic skin ulcer therapy in Jamaica. West Indian Med J. 2000 Mar;49(1):32-3. PMID 10786448
- [Background] Owoyele BV, Adebukola OM, Funmilayo AA, Soladoye AO. Anti-inflammatory activities of ethanolic extract of Carica papaya leaves. Inflammopharmacology. 2008 Aug;16(4):168-73. doi: 10.1007/s10787-008-7008-0. PMID 18759075
- [Background] Mahmood AA, Sihdik K, Salmah I. Wound healing activity of Carica papaya L. aqueous leaf extracts in rats. International Journal of Molecular Medicine and Advance Sciences 2005;1(4):398-401.
- [Background] Buensalido JS, Dimagiba TE. The efficacy and safety of 1.5% carica papaya latex cream compared to 2% ketoconazole cream and vehicle in the treatment of tinea corporis: A randomized, double blind, controlled trial. J Phil Dermatol Soc 2011 May;20(1):15-20.
- [Background] Canoy-Valencia H, King-Joanino SVB. An in vitro study of the therapeutic effects of Carica papaya against superficial pyodermas. Makati Medical Center Proceedings 1996;10:21-3.
- [Background] Ablang AMJ, Nuguid AS. In vitro activity of Carica papaya powdered extract alone and in combination with penicillin against clinical isolates of Streptococcus pyogenes. Makati Medical Center Proceedings 2000;14:11-5.
- [Background] Dawkins G, Hewitt H, Wint Y, Obiefuna PC, Wint B. Antibacterial effects of Carica papaya fruit on common wound organisms. West Indian Med J. 2003 Dec;52(4):290-2. PMID 15040064
- [Background] Doughari JH, Elmahmood AM, Manzara S. Studies on the antibacterial activity of root extracts of Carica papaya L. African Journal of Microbiology Research 2007 August:37-41.
- [Background] Okechukwu RI, Obasi KO, Nnoli MC, Ukaoma AA. Antimicrobial properties and preliminary phytochemical analysis of Carica papaya leaf. Advances in Science and Technology 2010;4(1):45-8.
- [Background] Suresh K, Deepa P, Harisaranraj R, Achudhan V. Antimicrobial and phytochemical investication of the Carica papaya L., Cynodon dactylon (L.) Pers., Euphorbia herta L. Melia azedarach L., and Psidium guajava L. Ethnobotanical Leaflets 2008;12:1184-91.
- [Background] Celis MA, Verallo-Rowell VM. Carica papaya versus Fucidin cream in the treatment of superficial pyodermas in pediatric patients: A double blind study. (Unpublished, 1996).
- [Background] Oduola T, Adeniyi FAA, Ogunyemi EO, Bello IS, Idowu TO, Subair HG. Toxicity studies on an unripe Carica papaya aqueous extract: biochemical and haematological effects in wistar albino rats. Journal of Medicinal Plants Research 2007 August;1(1):1-4.
- [Background] Iliev D, Elsner P. Generalized drug reaction due to papaya juice in throat lozenges. Dermatology. 1997;194(4):364-6. doi: 10.1159/000246142. PMID 9252760
- [Background] Niinimaki A, Reijula K, Pirila T, Koistinen AM. Papain-induced allergic rhinoconjunctivitis in a cosmetologist. J Allergy Clin Immunol. 1993 Sep;92(3):492-3. doi: 10.1016/0091-6749(93)90129-4. No abstract available. PMID 8360400